CLINICAL TRIAL: NCT06591663
Title: Can Cognitive Therapy Rating Scale (CTRS) be Used Across Cultures? Enhancing Cultural Relevance of CTRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PACTCTRS24
Record Dates: First submitted 2024-06-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- implementation of culturally adapted Urdu version of the Cognitive Therapy Rating Scale (CTRS) (Experimental)
  Interventions: Behavioral: Cognitive Therapy Rating Scale (CTRS)

INTERVENTIONS:
Behavioral: Cognitive Therapy Rating Scale (CTRS) — CBT is the Cognitive Therapy Rating Scale (CTRS), an important assessment tool designed to assess the quality and effectiveness of cognitive therapy sessions.
  Mental health professionals, such as therapists and psychologists, commonly use the CTRS to evaluate various aspects of a therapy session. This includes the extent to which the therapist adheres to CBT principles, their skill in applying cognitive and behavioral techniques, their ability to develop a therapeutic relationship with the client, and the overall quality of the session. The scale may also include specific criteria or items that another trained therapist or researcher observes based on their observations during the therapy session (Pingol, 2023).

SUMMARY:
Translate and adapt the Cognitive Therapy Rating Scale (CTRS) into Urdu language and establishing the psychometric properties (reliability, validity, and norms) of the translated scale

DETAILED DESCRIPTION:
The purpose of this study is to increase the accessibility and accuracy of clinical assessments, ultimately improving the quality of mental health care delivery and advancing research in the field of clinical psychology within Urdu-speaking communities

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 to 65 years At least 5 years of education Score of 8 or higher on Hospital Anxiety and Depression Scale-Depression or Anxiety scales as measured by their primary care clinician

Exclusion Criteria:

* Substance use disorder according to DSM-5 TR criteria Significant cognitive impairment (for example, profound learning disability or dementia) Active psychosis as determined by their primary care clinician

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-08 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Establishing the psychometric properties of the translated CTRS scale | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Association of Cognitive Therapists, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No